CLINICAL TRIAL: NCT02809833
Title: Tocilizumab for the Treatment of Rheumatoid Arthritis: Findings on The Use of Tocilizumab in Daily Clinical Routine
Brief Title: Use of Tocilizumab for Rheumatoid Arthritis (RA) in Daily Routine
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22734
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab for RA in Routine Practice: Participants from routine clinical practice in Germany who are receiving tocilizumab for RA according to SmPC are eligible.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab must be selected by the treating physician in advance of the study and will be not provided by the Sponsor. The dose/regimen are at the discretion of the prescriber. However, tocilizumab in the SmPC is specified as 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion at 4-week intervals.
  Other Names: Actemra/RoActemra

SUMMARY:
This prospective, multicenter, non-interventional study will enroll participants from routine clinical practice in Germany who are receiving tocilizumab for RA. The objective of the study is systematic collection of data on use of tocilizumab in daily routine with special emphasis on treatment decision by the prescriber, compliance with Summary of Product Characteristics (SmPC), and documentation of relevant activity scores and adverse drug reactions (ADRs). The maximum observation period will be 12 months per participant.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe RA
* Tocilizumab indicated in accordance with SmPC and chosen by the treating physician in advance of the study

Exclusion Criteria:

* None specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from routine clinical practice in Germany who are receiving tocilizumab for RA according to SmPC are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab for Rheumatoid Arthritis (RA) in Routine Practice: Participants from routine clinical practice in Germany who received tocilizumab for RA according to the Summary of Product Characteristics (SmPC) were observed for up to 12 months. Tocilizumab must have been selected by the treating physician in advance of the study and was not provided by the Sponsor. According to SmPC, tocilizumab was given as 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion at 4-week intervals.
Period: Overall Study
Arm/Group | Tocilizumab for Rheumatoid Arthritis (RA) in Routine Practice
Started | 850
Completed | 550
Not Completed | 300
Not completed — Death | 3
Not completed — Intolerance | 54
Not completed — Lack of Efficacy | 89
Not completed — Remission/Treatment No Longer Needed | 3
Not completed — Noncompliance | 1
Not completed — Withdrawal by Subject | 34
Not completed — Lost to Follow-up | 35
Not completed — Adverse Event (AE) | 24
Not completed — Other | 5
Not completed — Missing Information | 52

BASELINE CHARACTERISTICS:
Population: All Enrolled Population: All participants enrolled into the study.
Groups:
- Tocilizumab for RA in Routine Practice: Participants from routine clinical practice in Germany who received tocilizumab for RA according to SmPC were observed for up to 12 months. Tocilizumab must have been selected by the treating physician in advance of the study and was not provided by the Sponsor. According to SmPC, tocilizumab was given as 8 mg/kg via IV infusion at 4-week intervals.
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 640
  Male | 210

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Categorized Laboratory Data Available at Baseline
Description: SmPC recommendations were specified in the collection of routine laboratory samples for alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), absolute neutrophil count (ANC), and low platelet count to guide dose decisions. Laboratory values for ALAT and ASAT were to be categorized in reference to the institution-specific upper limit of normal (ULN). Laboratory values for ANC and platelet count were to be categorized in reference to a normal range outlined in the SmPC. This range was 0.5 to 1 × 10^9 cells per liter (cells/L) for ANC and 50 to 100 × 10^3 cells per microliter (cells/μL) for platelet count. The percentage of participants with greater than or equal to (≥) 1 documented/evaluable laboratory value at Baseline was reported, along with the percentage of participants with categorized laboratory data available for each individual parameter.
Time Frame: Baseline
Population: All Enrolled Population.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 850
percentage of participants
  ≥1 Documented/Evaluable Laboratory Value | 98.6
  ASAT Categorized | 49.2
  ALAT Categorized | 63.5
  ANC Categorized | 7.3
  Platelet Count Categorized | 82.9

2. Primary Outcome: Percentage of Participants With Categorized Laboratory Data Available at Week 24
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and low platelet count to guide dose decisions. Laboratory values for ALAT and ASAT were to be categorized in reference to the institution-specific ULN. Laboratory values for ANC and platelet count were to be categorized in reference to a normal range outlined in the SmPC. This range was 0.5 to 1 × 10^9 cells/L for ANC and 50 to 100 × 10^3 cells/μL for platelet count. The percentage of participants with ≥1 documented/evaluable laboratory value at Week 24 was reported, along with the percentage of participants with categorized laboratory data available for each individual parameter.
Time Frame: Week 24
Population: All Enrolled Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 598
percentage of participants
  ≥1 Documented/Evaluable Laboratory Value | 87.6
  ASAT Categorized | 31.6
  ALAT Categorized | 42.6
  ANC Categorized | 4.2
  Platelet Count Categorized | 58.9

3. Primary Outcome: Percentage of Participants With Categorized Laboratory Data Available at Week 52
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and low platelet count to guide dose decisions. Laboratory values for ALAT and ASAT were to be categorized in reference to the institution-specific ULN. Laboratory values for ANC and platelet count were to be categorized in reference to a normal range outlined in the SmPC. This range was 0.5 to 1 × 10^9 cells/L for ANC and 50 to 100 × 10^3 cells/μL for platelet count. The percentage of participants with ≥1 documented/evaluable laboratory value at Week 52 was reported, along with the percentage of participants with categorized laboratory data available for each individual parameter.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 551
percentage of participants
  ≥1 Documented/Evaluable Laboratory Value | 86.4
  ASAT Categorized | 29.0
  ALAT Categorized | 39.9
  ANC Categorized | 5.6
  Platelet Count Categorized | 60.1

4. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 4
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values greater than (>) 1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC less than (<) 0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 4.
Time Frame: Week 4
Population: All Enrolled Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for the endpoint. The number of participants who had available data for both the specific laboratory parameter and for the possible dose change at the corresponding visit (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 701
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=283) | 0.7
  ASAT: >1 to 3 × ULN, Adjustment: No (n=283) | 14.5
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=283) | 0.4
  ASAT: >1 to 3 × ULN, Interruption: No (n=283) | 14.8
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=283) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=283) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=283) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=283) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=283) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=283) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=283) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=283) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=371) | 0.5
  ALAT: >1 to 3 × ULN, Adjustment: No (n=371) | 23.2
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=371) | 0.5
  ALAT: >1 to 3 × ULN, Interruption: No (n=371) | 23.2
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=371) | 0.3
  ALAT: >3 to 5 × ULN, Adjustment: No (n=371) | 1.1
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=371) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=371) | 1.3
  ALAT: >5 × ULN, Adjustment: Yes (n=371) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=371) | 0.3
  ALAT: >5 × ULN, Interruption: Yes (n=371) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=371) | 0.3
  ANC: <0.5, Adjustment: Yes (n=46) | 0.0
  ANC: <0.5, Adjustment: No (n=46) | 0.0
  ANC: <0.5, Interruption: Yes (n=46) | 0.0
  ANC: <0.5, Interruption: No (n=46) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=46) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=46) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=46) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=46) | 0.0
  Platelets: <50, Adjustment: Yes (n=481) | 0.0
  Platelets: <50, Adjustment: No (n=481) | 0.0
  Platelets: <50, Interruption: Yes (n=481) | 0.0
  Platelets: <50, Interruption: No (n=481) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=481) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=481) | 0.2
  Platelets: 50 to 100, Interruption: Yes (n=481) | 0.0
  Platelets: 50 to 100, Interruption: No (n=481) | 0.2

5. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 8
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 8.
Time Frame: Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 629
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=242) | 0.0
  ASAT: >1 to 3 × ULN, Adjustment: No (n=242) | 13.2
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=243) | 0.8
  ASAT: >1 to 3 × ULN, Interruption: No (n=243) | 11.9
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=242) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=242) | 0.4
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=243) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=243) | 0.4
  ASAT: >5 × ULN, Adjustment: Yes (n=242) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=242) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=243) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=243) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=329) | 0.6
  ALAT: >1 to 3 × ULN, Adjustment: No (n=329) | 26.1
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=330) | 1.2
  ALAT: >1 to 3 × ULN, Interruption: No (n=330) | 25.2
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=329) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=329) | 1.2
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=330) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=330) | 1.2
  ALAT: >5 × ULN, Adjustment: Yes (n=329) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=329) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=330) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=330) | 0.0
  ANC: <0.5, Adjustment: Yes (n=41) | 0.0
  ANC: <0.5, Adjustment: No (n=41) | 0.0
  ANC: <0.5, Interruption: Yes (n=41) | 0.0
  ANC: <0.5, Interruption: No (n=41) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=41) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=41) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=41) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=41) | 0.0
  Platelets: <50, Adjustment: Yes (n=442) | 0.0
  Platelets: <50, Adjustment: No (n=442) | 0.0
  Platelets: <50, Interruption: Yes (n=443) | 0.0
  Platelets: <50, Interruption: No (n=443) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=442) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=442) | 0.5
  Platelets: 50 to 100, Interruption: Yes (n=443) | 0.0
  Platelets: 50 to 100, Interruption: No (n=443) | 0.5

6. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 12
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 12.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 574
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=229) | 0.0
  ASAT: >1 to 3 × ULN, Adjustment: No (n=229) | 18.3
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=230) | 1.3
  ASAT: >1 to 3 × ULN, Interruption: No (n=230) | 16.5
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=229) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=229) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=230) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=230) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=229) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=229) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=230) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=230) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=300) | 1.3
  ALAT: >1 to 3 × ULN, Adjustment: No (n=300) | 23.0
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=301) | 1.0
  ALAT: >1 to 3 × ULN, Interruption: No (n=301) | 22.9
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=300) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=300) | 1.3
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=301) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=301) | 1.3
  ALAT: >5 × ULN, Adjustment: Yes (n=300) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=300) | 0.3
  ALAT: >5 × ULN, Interruption: Yes (n=301) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=301) | 0.3
  ANC: <0.5, Adjustment: Yes (n=31) | 0.0
  ANC: <0.5, Adjustment: No (n=31) | 0.0
  ANC: <0.5, Interruption: Yes (n=31) | 0.0
  ANC: <0.5, Interruption: No (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=31) | 0.0
  Platelets: <50, Adjustment: Yes (n=410) | 0.0
  Platelets: <50, Adjustment: No (n=410) | 0.0
  Platelets: <50, Interruption: Yes (n=411) | 0.0
  Platelets: <50, Interruption: No (n=411) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=410) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=410) | 0.2
  Platelets: 50 to 100, Interruption: Yes (n=411) | 0.0
  Platelets: 50 to 100, Interruption: No (n=411) | 0.2

7. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 16
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 16.
Time Frame: Week 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 545
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=214) | 0.9
  ASAT: >1 to 3 × ULN, Adjustment: No (n=214) | 16.8
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=214) | 0.5
  ASAT: >1 to 3 × ULN, Interruption: No (n=214) | 16.8
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=214) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=214) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=214) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=214) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=214) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=214) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=214) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=214) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=282) | 1.4
  ALAT: >1 to 3 × ULN, Adjustment: No (n=282) | 23.4
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=282) | 0.4
  ALAT: >1 to 3 × ULN, Interruption: No (n=282) | 24.1
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=282) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=282) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=282) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=282) | 0.0
  ALAT: >5 × ULN, Adjustment: Yes (n=282) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=282) | 0.4
  ALAT: >5 × ULN, Interruption: Yes (n=282) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=282) | 0.4
  ANC: <0.5, Adjustment: Yes (n=31) | 0.0
  ANC: <0.5, Adjustment: No (n=31) | 0.0
  ANC: <0.5, Interruption: Yes (n=31) | 0.0
  ANC: <0.5, Interruption: No (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=31) | 0.0
  Platelets: <50, Adjustment: Yes (n=378) | 0.0
  Platelets: <50, Adjustment: No (n=378) | 0.0
  Platelets: <50, Interruption: Yes (n=378) | 0.0
  Platelets: <50, Interruption: No (n=378) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=378) | 0.3
  Platelets: 50 to 100, Adjustment: No (n=378) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=378) | 0.0
  Platelets: 50 to 100, Interruption: No (n=378) | 0.5

8. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 20
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 20.
Time Frame: Week 20
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 518
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=175) | 0.6
  ASAT: >1 to 3 × ULN, Adjustment: No (n=175) | 18.9
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=175) | 1.1
  ASAT: >1 to 3 × ULN, Interruption: No (n=175) | 18.3
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=175) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=175) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=175) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=175) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=175) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=175) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=175) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=175) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=253) | 0.8
  ALAT: >1 to 3 × ULN, Adjustment: No (n=253) | 23.3
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=253) | 0.8
  ALAT: >1 to 3 × ULN, Interruption: No (n=253) | 23.3
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=253) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=253) | 1.6
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=253) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=253) | 1.6
  ALAT: >5 × ULN, Adjustment: Yes (n=253) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=253) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=253) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=253) | 0.0
  ANC: <0.5, Adjustment: Yes (n=31) | 0.0
  ANC: <0.5, Adjustment: No (n=31) | 3.2
  ANC: <0.5, Interruption: Yes (n=31) | 0.0
  ANC: <0.5, Interruption: No (n=31) | 3.2
  ANC: 0.5 to 1, Adjustment: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=31) | 0.0
  Platelets: <50, Adjustment: Yes (n=352) | 0.0
  Platelets: <50, Adjustment: No (n=352) | 0.0
  Platelets: <50, Interruption: Yes (n=352) | 0.0
  Platelets: <50, Interruption: No (n=352) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=352) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=352) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=352) | 0.0
  Platelets: 50 to 100, Interruption: No (n=352) | 0.3

9. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 24
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 24.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 524
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=189) | 0.5
  ASAT: >1 to 3 × ULN, Adjustment: No (n=189) | 15.9
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=189) | 0.0
  ASAT: >1 to 3 × ULN, Interruption: No (n=189) | 16.4
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=189) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=189) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=189) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=189) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=189) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=189) | 0.5
  ASAT: >5 × ULN, Interruption: Yes (n=189) | 0.5
  ASAT: >5 × ULN, Interruption: No (n=189) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=255) | 0.8
  ALAT: >1 to 3 × ULN, Adjustment: No (n=255) | 26.7
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=255) | 1.2
  ALAT: >1 to 3 × ULN, Interruption: No (n=255) | 25.9
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=255) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=255) | 0.4
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=255) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=255) | 0.4
  ALAT: >5 × ULN, Adjustment: Yes (n=255) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=255) | 0.4
  ALAT: >5 × ULN, Interruption: Yes (n=255) | 0.4
  ALAT: >5 × ULN, Interruption: No (n=255) | 0.0
  ANC: <0.5, Adjustment: Yes (n=25) | 0.0
  ANC: <0.5, Adjustment: No (n=25) | 0.0
  ANC: <0.5, Interruption: Yes (n=25) | 0.0
  ANC: <0.5, Interruption: No (n=25) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=25) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=25) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=25) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=25) | 0.0
  Platelets: <50, Adjustment: Yes (n=350) | 0.0
  Platelets: <50, Adjustment: No (n=350) | 0.0
  Platelets: <50, Interruption: Yes (n=352) | 0.0
  Platelets: <50, Interruption: No (n=352) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=350) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=350) | 0.9
  Platelets: 50 to 100, Interruption: Yes (n=352) | 0.0
  Platelets: 50 to 100, Interruption: No (n=352) | 0.9

10. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 28
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 28.
Time Frame: Week 28
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 471
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=173) | 0.0
  ASAT: >1 to 3 × ULN, Adjustment: No (n=173) | 15.6
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=173) | 0.6
  ASAT: >1 to 3 × ULN, Interruption: No (n=173) | 15.0
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=173) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=173) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=173) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=173) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=173) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=173) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=173) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=173) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=233) | 0.9
  ALAT: >1 to 3 × ULN, Adjustment: No (n=233) | 21.5
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=233) | 1.3
  ALAT: >1 to 3 × ULN, Interruption: No (n=233) | 21.0
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=233) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=233) | 1.3
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=233) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=233) | 1.3
  ALAT: >5 × ULN, Adjustment: Yes (n=233) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=233) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=233) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=233) | 0.0
  ANC: <0.5, Adjustment: Yes (n=28) | 0.0
  ANC: <0.5, Adjustment: No (n=28) | 0.0
  ANC: <0.5, Interruption: Yes (n=28) | 0.0
  ANC: <0.5, Interruption: No (n=28) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=28) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=28) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=28) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=28) | 0.0
  Platelets: <50, Adjustment: Yes (n=333) | 0.0
  Platelets: <50, Adjustment: No (n=333) | 0.0
  Platelets: <50, Interruption: Yes (n=333) | 0.0
  Platelets: <50, Interruption: No (n=333) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=333) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=333) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=333) | 0.0
  Platelets: 50 to 100, Interruption: No (n=333) | 0.3

11. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 32
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 32.
Time Frame: Week 32
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 473
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=163) | 1.2
  ASAT: >1 to 3 × ULN, Adjustment: No (n=163) | 12.3
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=163) | 0.6
  ASAT: >1 to 3 × ULN, Interruption: No (n=163) | 12.9
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=163) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=163) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=163) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=163) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=163) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=163) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=163) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=163) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=225) | 1.3
  ALAT: >1 to 3 × ULN, Adjustment: No (n=225) | 21.8
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=225) | 0.4
  ALAT: >1 to 3 × ULN, Interruption: No (n=225) | 22.7
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=225) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=225) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=225) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=225) | 0.0
  ALAT: >5 × ULN, Adjustment: Yes (n=225) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=225) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=225) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=225) | 0.0
  ANC: <0.5, Adjustment: Yes (n=26) | 0.0
  ANC: <0.5, Adjustment: No (n=26) | 0.0
  ANC: <0.5, Interruption: Yes (n=26) | 0.0
  ANC: <0.5, Interruption: No (n=26) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=26) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=26) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=26) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=26) | 0.0
  Platelets: <50, Adjustment: Yes (n=309) | 0.0
  Platelets: <50, Adjustment: No (n=309) | 0.0
  Platelets: <50, Interruption: Yes (n=309) | 0.0
  Platelets: <50, Interruption: No (n=309) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=309) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=309) | 0.6
  Platelets: 50 to 100, Interruption: Yes (n=309) | 0.0
  Platelets: 50 to 100, Interruption: No (n=309) | 0.6

12. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 36
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 36.
Time Frame: Week 36
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 421
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=143) | 0.7
  ASAT: >1 to 3 × ULN, Adjustment: No (n=143) | 19.6
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=143) | 0.0
  ASAT: >1 to 3 × ULN, Interruption: No (n=143) | 20.3
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=143) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=143) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=143) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=143) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=143) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=143) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=143) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=143) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=194) | 1.5
  ALAT: >1 to 3 × ULN, Adjustment: No (n=194) | 23.2
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=194) | 0.5
  ALAT: >1 to 3 × ULN, Interruption: No (n=194) | 24.2
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=194) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=194) | 0.5
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=194) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=194) | 0.5
  ALAT: >5 × ULN, Adjustment: Yes (n=194) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=194) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=194) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=194) | 0.0
  ANC: <0.5, Adjustment: Yes (n=25) | 0.0
  ANC: <0.5, Adjustment: No (n=25) | 0.0
  ANC: <0.5, Interruption: Yes (n=25) | 0.0
  ANC: <0.5, Interruption: No (n=25) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=25) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=25) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=25) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=25) | 0.0
  Platelets: <50, Adjustment: Yes (n=282) | 0.0
  Platelets: <50, Adjustment: No (n=282) | 0.0
  Platelets: <50, Interruption: Yes (n=282) | 0.0
  Platelets: <50, Interruption: No (n=282) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=282) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=282) | 1.1
  Platelets: 50 to 100, Interruption: Yes (n=282) | 0.0
  Platelets: 50 to 100, Interruption: No (n=282) | 1.1

13. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 40
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 40.
Time Frame: Week 40
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 434
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=138) | 0.0
  ASAT: >1 to 3 × ULN, Adjustment: No (n=138) | 20.3
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=138) | 0.0
  ASAT: >1 to 3 × ULN, Interruption: No (n=138) | 20.3
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=138) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=138) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=138) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=138) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=138) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=138) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=138) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=138) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=202) | 0.5
  ALAT: >1 to 3 × ULN, Adjustment: No (n=202) | 21.3
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=202) | 0.0
  ALAT: >1 to 3 × ULN, Interruption: No (n=202) | 21.8
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=202) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=202) | 0.5
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=202) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=202) | 0.5
  ALAT: >5 × ULN, Adjustment: Yes (n=202) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=202) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=202) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=202) | 0.0
  ANC: <0.5, Adjustment: Yes (n=22) | 0.0
  ANC: <0.5, Adjustment: No (n=22) | 0.0
  ANC: <0.5, Interruption: Yes (n=22) | 0.0
  ANC: <0.5, Interruption: No (n=22) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=22) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=22) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=22) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=22) | 0.0
  Platelets: <50, Adjustment: Yes (n=296) | 0.0
  Platelets: <50, Adjustment: No (n=296) | 0.0
  Platelets: <50, Interruption: Yes (n=296) | 0.0
  Platelets: <50, Interruption: No (n=296) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=296) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=296) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=296) | 0.0
  Platelets: 50 to 100, Interruption: No (n=296) | 0.3

14. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 44
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 44.
Time Frame: Week 44
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 415
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=140) | 0.7
  ASAT: >1 to 3 × ULN, Adjustment: No (n=140) | 15.7
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=140) | 0.0
  ASAT: >1 to 3 × ULN, Interruption: No (n=140) | 16.4
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=140) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=140) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=140) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=140) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=140) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=140) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=140) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=140) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=197) | 1.5
  ALAT: >1 to 3 × ULN, Adjustment: No (n=197) | 24.4
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=197) | 0.5
  ALAT: >1 to 3 × ULN, Interruption: No (n=197) | 24.9
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=197) | 0.0
  ALAT: >3 to 5 × ULN, Adjustment: No (n=197) | 0.5
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=197) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=197) | 0.5
  ALAT: >5 × ULN, Adjustment: Yes (n=197) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=197) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=197) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=197) | 0.0
  ANC: <0.5, Adjustment: Yes (n=26) | 0.0
  ANC: <0.5, Adjustment: No (n=26) | 0.0
  ANC: <0.5, Interruption: Yes (n=26) | 0.0
  ANC: <0.5, Interruption: No (n=26) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=26) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=26) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=26) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=26) | 0.0
  Platelets: <50, Adjustment: Yes (n=279) | 0.0
  Platelets: <50, Adjustment: No (n=279) | 0.0
  Platelets: <50, Interruption: Yes (n=279) | 0.0
  Platelets: <50, Interruption: No (n=279) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=279) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=279) | 0.4
  Platelets: 50 to 100, Interruption: Yes (n=279) | 0.0
  Platelets: 50 to 100, Interruption: No (n=279) | 0.4

15. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 48
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 48.
Time Frame: Week 48
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 414
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=130) | 1.5
  ASAT: >1 to 3 × ULN, Adjustment: No (n=130) | 16.2
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=131) | 0.0
  ASAT: >1 to 3 × ULN, Interruption: No (n=131) | 17.6
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=130) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=130) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=131) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=131) | 0.0
  ASAT: >5 × ULN, Adjustment: Yes (n=130) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=130) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=131) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=131) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=190) | 1.1
  ALAT: >1 to 3 × ULN, Adjustment: No (n=190) | 21.6
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=191) | 0.5
  ALAT: >1 to 3 × ULN, Interruption: No (n=191) | 22.0
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=190) | 0.5
  ALAT: >3 to 5 × ULN, Adjustment: No (n=190) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=191) | 0.0
  ALAT: >3 to 5 × ULN, Interruption: No (n=191) | 0.5
  ALAT: >5 × ULN, Adjustment: Yes (n=190) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=190) | 0.0
  ALAT: >5 × ULN, Interruption: Yes (n=191) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=191) | 0.0
  ANC: <0.5, Adjustment: Yes (n=22) | 0.0
  ANC: <0.5, Adjustment: No (n=22) | 0.0
  ANC: <0.5, Interruption: Yes (n=22) | 0.0
  ANC: <0.5, Interruption: No (n=22) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=22) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=22) | 4.5
  ANC: 0.5 to 1, Interruption: Yes (n=22) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=22) | 4.5
  Platelets: <50, Adjustment: Yes (n=286) | 0.0
  Platelets: <50, Adjustment: No (n=286) | 0.0
  Platelets: <50, Interruption: Yes (n=287) | 0.0
  Platelets: <50, Interruption: No (n=287) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=286) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=286) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=287) | 0.0
  Platelets: 50 to 100, Interruption: No (n=287) | 0.3

16. Primary Outcome: Percentage of Participants With or Without Tocilizumab Dose Adjustment or Interruption at Week 52
Description: SmPC recommendations were specified in the collection of routine laboratory samples for ALAT, ASAT, ANC, and platelet count to guide dose decisions. Dose adjustment was recommended in response to ALAT/ASAT values >1 to 3 × ULN. Dose interruption was recommended in response to ALAT/ASAT values >3 to 5 × ULN, ANC of 0.5 to 1 × 10^9 cells/L, or platelet count of 50 to 100 × 10^3 cells/μL, until the values returned to acceptable ranges as per the SmPC. Discontinuation of tocilizumab was recommended for any ALAT/ASAT values >5 × ULN, ANC <0.5 × 10^9 cells/L, or platelet count <50 × 10^3 cells/μL. The percentage of participants from each laboratory value category with ("Yes") or without ("No") tocilizumab dose adjustment or interruption was reported at Week 52.
Time Frame: Week 52
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 476
percentage of participants
  ASAT: >1 to 3 × ULN, Adjustment: Yes (n=160) | 1.9
  ASAT: >1 to 3 × ULN, Adjustment: No (n=160) | 18.1
  ASAT: >1 to 3 × ULN, Interruption: Yes (n=160) | 2.5
  ASAT: >1 to 3 × ULN, Interruption: No (n=160) | 17.5
  ASAT: >3 to 5 × ULN, Adjustment: Yes (n=160) | 0.0
  ASAT: >3 to 5 × ULN, Adjustment: No (n=160) | 0.6
  ASAT: >3 to 5 × ULN, Interruption: Yes (n=160) | 0.0
  ASAT: >3 to 5 × ULN, Interruption: No (n=160) | 0.6
  ASAT: >5 × ULN, Adjustment: Yes (n=160) | 0.0
  ASAT: >5 × ULN, Adjustment: No (n=160) | 0.0
  ASAT: >5 × ULN, Interruption: Yes (n=160) | 0.0
  ASAT: >5 × ULN, Interruption: No (n=160) | 0.0
  ALAT: >1 to 3 × ULN, Adjustment: Yes (n=220) | 3.2
  ALAT: >1 to 3 × ULN, Adjustment: No (n=220) | 22.7
  ALAT: >1 to 3 × ULN, Interruption: Yes (n=220) | 1.4
  ALAT: >1 to 3 × ULN, Interruption: No (n=220) | 24.1
  ALAT: >3 to 5 × ULN, Adjustment: Yes (n=220) | 0.5
  ALAT: >3 to 5 × ULN, Adjustment: No (n=220) | 2.3
  ALAT: >3 to 5 × ULN, Interruption: Yes (n=220) | 0.5
  ALAT: >3 to 5 × ULN, Interruption: No (n=220) | 2.3
  ALAT: >5 × ULN, Adjustment: Yes (n=220) | 0.0
  ALAT: >5 × ULN, Adjustment: No (n=220) | 0.5
  ALAT: >5 × ULN, Interruption: Yes (n=220) | 0.0
  ALAT: >5 × ULN, Interruption: No (n=220) | 0.5
  ANC: <0.5, Adjustment: Yes (n=31) | 0.0
  ANC: <0.5, Adjustment: No (n=31) | 0.0
  ANC: <0.5, Interruption: Yes (n=31) | 0.0
  ANC: <0.5, Interruption: No (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Adjustment: No (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: Yes (n=31) | 0.0
  ANC: 0.5 to 1, Interruption: No (n=31) | 0.0
  Platelets: <50, Adjustment: Yes (n=331) | 0.0
  Platelets: <50, Adjustment: No (n=331) | 0.0
  Platelets: <50, Interruption: Yes (n=331) | 0.0
  Platelets: <50, Interruption: No (n=331) | 0.0
  Platelets: 50 to 100, Adjustment: Yes (n=331) | 0.0
  Platelets: 50 to 100, Adjustment: No (n=331) | 0.3
  Platelets: 50 to 100, Interruption: Yes (n=331) | 0.0
  Platelets: 50 to 100, Interruption: No (n=331) | 0.3

17. Primary Outcome: Percentage of Participants With Tocilizumab Dose Adjustments by Reason
Description: The percentage of participants with any tocilizumab dose adjustment during the study was reported among all reasons given for tocilizumab dose adjustments, as provided in the CRF. The sum of all reasons may add up to >100 percent (%) because more than one reason could be given for each dose change. In the table presented, "Other Reasons" refers to any reason other than those specified in categories. Similarly, "Other Laboratory Change" refers to a change in any laboratory parameter other than those specified in categories.
Time Frame: Baseline to end of treatment (up to 12 months)
Population: All Enrolled Population. The "Number of Participants Analyzed" reflects the number of participants who had at least one tocilizumab dose adjustment during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 199
percentage of participants
  Weight Change | 54.3
  Adverse Event/Non-RA Medical Cause | 11.1
  Remission/RA Improvement | 10.6
  Maximum Dose per SmPC | 9.0
  RA Activity | 8.5
  Dose Titration | 6.5
  Other Reasons | 5.5
  Participant Request | 4.5
  Liver Enzyme Laboratory Change | 4.0
  Neutrophil Laboratory Change | 1.5
  Platelet Laboratory Change | 0.5
  Other Laboratory Change | 4.5
  Not Specified Laboratory Change | 0.5

18. Primary Outcome: 28-Joint Disease Activity Score (DAS28) at Baseline
Description: The DAS28 was derived from assessments of erythrocyte sedimentation rate (ESR), tender joint count (TJC), swollen joint count (SJC), and general health according to 100-millimeter (mm) Visual Analog Scale (VAS). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in millimeters per hour (mm/h). DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The score at Baseline was reported.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 728
units on a scale | 5.5 (1.3)

19. Primary Outcome: Change in DAS28 From Baseline to Week 4
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 4 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 516
units on a scale | -1.8 (1.4)

20. Primary Outcome: Change in DAS28 From Baseline to Week 8
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 8 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 453
units on a scale | -2.3 (1.5)

21. Primary Outcome: Change in DAS28 From Baseline to Week 12
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 12 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 424
units on a scale | -2.4 (1.6)

22. Primary Outcome: Change in DAS28 From Baseline to Week 16
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 16 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 392
units on a scale | -2.6 (1.6)

23. Primary Outcome: Change in DAS28 From Baseline to Week 20
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 20 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 389
units on a scale | -2.6 (1.6)

24. Primary Outcome: Change in DAS28 From Baseline to Week 24
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 24 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 389
units on a scale | -2.7 (1.6)

25. Primary Outcome: Change in DAS28 From Baseline to Week 28
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 28 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 341
units on a scale | -2.7 (1.6)

26. Primary Outcome: Change in DAS28 From Baseline to Week 32
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 32 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 356
units on a scale | -2.8 (1.5)

27. Primary Outcome: Change in DAS28 From Baseline to Week 36
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 36 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 312
units on a scale | -2.9 (1.7)

28. Primary Outcome: Change in DAS28 From Baseline to Week 40
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 40 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 40
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 326
units on a scale | -2.8 (1.7)

29. Primary Outcome: Change in DAS28 From Baseline to Week 44
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 44 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 305
units on a scale | -3.0 (1.6)

30. Primary Outcome: Change in DAS28 From Baseline to Week 48
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 48 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 316
units on a scale | -2.9 (1.7)

31. Primary Outcome: Change in DAS28 From Baseline to Week 52
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 52 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 353
units on a scale | -2.9 (1.7)

32. Primary Outcome: TJC at Baseline
Description: A total of 28 joints were assessed for tenderness. The number of tender joints at Baseline was reported and could range from 0 to 28, where higher values represented more tender joints.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 823
tender joints | 9.5 (6.7)

33. Primary Outcome: Change in TJC From Baseline to Week 12
Description: A total of 28 joints were assessed for tenderness. The number of tender joints could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to Week 12 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 593
tender joints | -5.2 (6.3)

34. Primary Outcome: Change in TJC From Baseline to Week 24
Description: A total of 28 joints were assessed for tenderness. The number of tender joints could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to Week 24 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 540
tender joints | -6.2 (7.0)

35. Primary Outcome: Change in TJC From Baseline to Week 36
Description: A total of 28 joints were assessed for tenderness. The number of tender joints could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to Week 36 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 446
tender joints | -6.6 (6.8)

36. Primary Outcome: Change in TJC From Baseline to Week 52
Description: A total of 28 joints were assessed for tenderness. The number of tender joints could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to Week 52 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 492
tender joints | -6.7 (6.9)

37. Primary Outcome: SJC at Baseline
Description: A total of 28 joints were assessed for swollenness. The number of swollen joints at Baseline was reported and could range from 0 to 28, where higher values represented more swollen joints.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 829
swollen joints | 8.1 (6.0)

38. Primary Outcome: Change in SJC From Baseline to Week 12
Description: A total of 28 joints were assessed for swollenness. The number of swollen joints could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to Week 12 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 600
swollen joints | -4.6 (5.7)

39. Primary Outcome: Change in SJC From Baseline to Week 24
Description: A total of 28 joints were assessed for swollenness. The number of swollen joints could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to Week 24 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 545
swollen joints | -5.2 (5.9)

40. Primary Outcome: Change in SJC From Baseline to Week 36
Description: A total of 28 joints were assessed for swollenness. The number of swollen joints could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to Week 36 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 446
swollen joints | -6.0 (6.1)

41. Primary Outcome: Change in SJC From Baseline to Week 52
Description: A total of 28 joints were assessed for swollenness. The number of swollen joints could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to Week 52 was reported, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 496
swollen joints | -6.0 (6.0)

42. Primary Outcome: VAS Score of Participant-Assessed Disease Activity at Baseline
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The VAS score at Baseline was reported.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 821
mm | 66.8 (20.0)

43. Primary Outcome: Change in VAS Score of Participant-Assessed Disease Activity From Baseline to Week 12
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 12 was reported, where negative changes indicated a decrease in participant-assessed disease activity.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 611
mm | -28.0 (25.0)

44. Primary Outcome: Change in VAS Score of Participant-Assessed Disease Activity From Baseline to Week 24
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 24 was reported, where negative changes indicated a decrease in participant-assessed disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 558
mm | -32.0 (25.5)

45. Primary Outcome: Change in VAS Score of Participant-Assessed Disease Activity From Baseline to Week 36
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 36 was reported, where negative changes indicated a decrease in participant-assessed disease activity.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 461
mm | -36.0 (27.2)

46. Primary Outcome: Change in VAS Score of Participant-Assessed Disease Activity From Baseline to Week 52
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 52 was reported, where negative changes indicated a decrease in participant-assessed disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 515
mm | -36.4 (26.8)

47. Primary Outcome: VAS Score of Physician-Assessed Disease Activity at Baseline
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The VAS score at Baseline was reported.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 819
mm | 62.7 (18.6)

48. Primary Outcome: Change in VAS Score of Physician-Assessed Disease Activity From Baseline to Week 12
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 12 was reported, where negative changes indicated a decrease in physician-assessed disease activity.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 605
mm | -29.6 (23.3)

49. Primary Outcome: Change in VAS Score of Physician-Assessed Disease Activity From Baseline to Week 24
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 24 was reported, where negative changes indicated a decrease in physician-assessed disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 552
mm | -34.5 (23.7)

50. Primary Outcome: Change in VAS Score of Physician-Assessed Disease Activity From Baseline to Week 36
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 36 was reported, where negative changes indicated a decrease in physician-assessed disease activity.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 455
mm | -37.3 (25.1)

51. Primary Outcome: Change in VAS Score of Physician-Assessed Disease Activity From Baseline to Week 52
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity. Higher scores corresponded to increased disease activity (0 mm = no disease activity and 100 mm = maximum disease activity). The change from Baseline to Week 52 was reported, where negative changes indicated a decrease in physician-assessed disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 513
mm | -38.5 (25.3)

52. Primary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 4
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the Week 4 visit and the DAS28 change from Baseline to Week 4. Participants with a score less than or equal to (≤) 3.2 and reduction of >1.2 points were assessed as having a "Good" response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a "Moderate" response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as non-responders with response recorded as "No Improvement".
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 516
percentage of participants
  Good | 31.8
  Moderate | 44.2
  No Improvement | 24.0

53. Primary Outcome: Percentage of Participants With EULAR Response at Week 12
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the Week 12 visit and the DAS28 change from Baseline to Week 12. Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a "Good" response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a "Moderate" response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as non-responders with response recorded as "No Improvement".
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 424
percentage of participants
  Good | 50.0
  Moderate | 36.3
  No Improvement | 13.7

54. Primary Outcome: Percentage of Participants With EULAR Response at Week 24
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the Week 24 visit and the DAS28 change from Baseline to Week 24. Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a "Good" response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a "Moderate" response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as non-responders with response recorded as "No Improvement".
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 389
percentage of participants
  Good | 54.8
  Moderate | 33.2
  No Improvement | 12.1

55. Primary Outcome: Percentage of Participants With EULAR Response at Week 36
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the Week 36 visit and the DAS28 change from Baseline to Week 36. Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a "Good" response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a "Moderate" response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as non-responders with response recorded as "No Improvement".
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 312
percentage of participants
  Good | 60.3
  Moderate | 28.5
  No Improvement | 11.2

56. Primary Outcome: Percentage of Participants With EULAR Response at Week 52
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the Week 52 visit and the DAS28 change from Baseline to Week 52. Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a "Good" response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a "Moderate" response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as non-responders with response recorded as "No Improvement".
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 353
percentage of participants
  Good | 62.3
  Moderate | 26.6
  No Improvement | 11.0

57. Primary Outcome: Percentage of Participants With Low Disease Activity Score (LDAS) According to DAS28 at Baseline
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. LDAS was defined as a DAS28 score ≤3.2 at Baseline.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 728
percentage of participants | 5.1

58. Primary Outcome: Percentage of Participants With LDAS According to DAS28 at Week 12
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. LDAS was defined as a DAS28 score ≤3.2 at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 459
percentage of participants | 55.1

59. Primary Outcome: Percentage of Participants With LDAS According to DAS28 at Week 24
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. LDAS was defined as a DAS28 score ≤3.2 at Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 427
percentage of participants | 59.3

60. Primary Outcome: Percentage of Participants With LDAS According to DAS28 at Week 36
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. LDAS was defined as a DAS28 score ≤3.2 at Week 36.
Time Frame: Week 36
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 349
percentage of participants | 65.3

61. Primary Outcome: Percentage of Participants With LDAS According to DAS28 at Week 52
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. LDAS was defined as a DAS28 score ≤3.2 at Week 52.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 396
percentage of participants | 66.4

62. Primary Outcome: Percentage of Participants With Remission According to DAS28 at Baseline
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Remission was defined as a DAS28 score <2.6 at Baseline.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 728
percentage of participants | 2.5

63. Primary Outcome: Percentage of Participants With Remission According to DAS28 at Week 12
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Remission was defined as a DAS28 score <2.6 at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 459
percentage of participants | 41.8

64. Primary Outcome: Percentage of Participants With Remission According to DAS28 at Week 24
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Remission was defined as a DAS28 score <2.6 at Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 427
percentage of participants | 45.7

65. Primary Outcome: Percentage of Participants With Remission According to DAS28 at Week 36
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Remission was defined as a DAS28 score <2.6 at Week 36.
Time Frame: Week 36
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 349
percentage of participants | 52.4

66. Primary Outcome: Percentage of Participants With Remission According to DAS28 at Week 52
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Remission was defined as a DAS28 score <2.6 at Week 52.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 396
percentage of participants | 55.1

67. Primary Outcome: Percentage of Participants With Minimum Clinically Important Improvement (MCII) According to DAS28 at Week 12
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. MCII was defined as DAS28 reduction of ≥1.2 points from Baseline to Week 12.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 424
percentage of participants | 76.7

68. Primary Outcome: Percentage of Participants With MCII According to DAS28 at Week 24
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. MCII was defined as DAS28 reduction of ≥1.2 points from Baseline to Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 389
percentage of participants | 82.0

69. Primary Outcome: Percentage of Participants With MCII According to DAS28 at Week 36
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. MCII was defined as DAS28 reduction of ≥1.2 points from Baseline to Week 36.
Time Frame: Baseline to Week 36
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 312
percentage of participants | 84.0

70. Primary Outcome: Percentage of Participants With MCII According to DAS28 at Week 52
Description: The DAS28 was derived from assessments of ESR, TJC, SJC, and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of tender joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. MCII was defined as DAS28 reduction of ≥1.2 points from Baseline to Week 52.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 353
percentage of participants | 84.7

71. Secondary Outcome: Percentage of Participants With AEs Considered Causally Related to Tocilizumab
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease associated with the use of tocilizumab. Worsened pre-existing conditions and laboratory or clinical tests that resulted in change or discontinuation of treatment were reported as AEs. The percentage of participants with treatment-related AEs (also known as adverse drug reactions) was reported as a separate endpoint and included both serious and non-serious AEs. Those AEs with a causal relationship reported as "definite", "probably", "possible", or "unlikely" were considered to be related to tocilizumab. If the causal relationship was reported as "unrelated", the AE was considered not related to tocilizumab treatment. Terms were reported verbatim as coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 12.0. The most common treatment-related AEs were reported, using those from the 10 highest incidence rate levels.
Time Frame: Baseline to end of treatment (up to 12 months)
Population: All Enrolled Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab for RA in Routine Practice
Number analyzed (Participants) | 850
percentage of participants
  Any Treatment-Related AE | 39.4
  Bronchitis | 3.4
  Nasopharyngitis | 2.9
  Pruritus | 2.4
  Headache | 2.1
  Hypercholesterolaemia | 1.9
  Diarrhoea | 1.4
  Hypertension | 1.4
  Respiratory tract infection | 1.4
  Sinusitis | 1.4
  Leukopenia | 1.3
  Nausea | 1.3
  Rash | 1.2
  Alopecia | 1.2
  Gamma-glutamyltransferase increased | 1.2
  Herpes zoster | 1.2
  Dizziness | 1.1
  Cystitis | 0.9
  Liver function test abnormal | 0.9
  Oral herpes | 0.9
  Upper respiratory tract infection | 0.9
  Urinary tract infection | 0.9

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (up to 12 months); assessed at Baseline and Weeks 4-8, 12-16, 20-24, 36, 52; assessments were also possible/optional at 4-week intervals between Baseline and Week 52
Description: Analysis Population Description: All Enrolled Population. Participants were asked about AEs at each study visit.
Arm/Group | Tocilizumab for RA in Routine Practice
Serious Adverse Events (participants affected / at risk) | 104/850
Other Adverse Events (participants affected / at risk) | 320/850
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab for RA in Routine Practice (N=850)
Anaemia (Blood and lymphatic system disorders) | 2
Bone marrow toxicity (Blood and lymphatic system disorders) | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Diplopia (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Anorectal varices haemorrhage (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Foreign body reaction (General disorders) | 1
General physical health deterioration (General disorders) | 2
Impaired healing (General disorders) | 2
Influenza like illness (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Ulcer (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 7
Bronchopneumonia (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 3
Gangrene (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Infection (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Post procedural infection (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone fistula (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Breast cyst excision (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Aortic thrombosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3
Iliac artery stenosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab for RA in Routine Practice (N=850)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 3
Tachycardia paroxysmal (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Eustachian tube disorder (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival cyst (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 3
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eczema eyelids (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Sicca syndrome (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Visual impairment (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Aphthous stomatitis (Gastrointestinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 14
Diverticulum (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Oesophageal discomfort (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 5
Retching (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 1
Chills (General disorders) | 2
Condition aggravated (General disorders) | 3
Drug ineffective (General disorders) | 2
Drug intolerance (General disorders) | 1
Fatigue (General disorders) | 7
Impaired healing (General disorders) | 4
Inflammation (General disorders) | 1
Infusion site erythema (General disorders) | 1
Infusion site pruritus (General disorders) | 1
Malaise (General disorders) | 2
Mucosa vesicle (General disorders) | 1
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 3
Borrelia infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 27
Bronchitis bacterial (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Cystitis (Infections and infestations) | 7
Erysipelas (Infections and infestations) | 5
Erysipeloid (Infections and infestations) | 1
Erythema migrans (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis norovirus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 2
Herpes simplex (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 7
Hordeolum (Infections and infestations) | 2
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 3
Lobar pneumonia (Infections and infestations) | 1
Localised infection (Infections and infestations) | 3
Measles (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 28
Onychomycosis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 7
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 3
Paronychia (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 14
Respiratory tract infection viral (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 7
Salmonellosis (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 9
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 5
Tooth abscess (Infections and infestations) | 2
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 7
Viral infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 4
Blood creatinine increased (Investigations) | 3
Blood pressure increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 2
C-reactive protein abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 9
Haemoglobin abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 3
Intraocular pressure increased (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Liver function test abnormal (Investigations) | 8
Low density lipoprotein increased (Investigations) | 2
Lymphocyte percentage increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Rheumatoid factor increased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Transaminases increased (Investigations) | 7
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 6
White blood cell count increased (Investigations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 9
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Migraine (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Polyneuropathy (Nervous system disorders) | 2
Post herpetic neuralgia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Bladder irritation (Renal and urinary disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10
Blood blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 6
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 17
Psoriasis (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 9
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Skin warm (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Menopause (Social circumstances) | 1
Arthrodesis (Surgical and medical procedures) | 2
Cataract operation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Haemorrhoid operation (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Shoulder arthroplasty (Surgical and medical procedures) | 1
Toe amputation (Surgical and medical procedures) | 1
Blood pressure fluctuation (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 13
Hypertensive crisis (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.